CLINICAL TRIAL: NCT02611843
Title: Peer Supported Web-based CBT for OEF/OIF Veterans With PTSD and Substance Misuse
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Syracuse VA Medical Center (U.S. Federal Agency)
Collaborators: National Development and Research Institutes, Inc. (Other)
Responsible Party: Principal Investigator, Kyle Possemato, Associate Director for Research, Center for Integrated Healthcare, Syracuse VA Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 487
Record Dates: First submitted 2015-11-19; First posted 2015-11-23 (Estimated); Last update posted 2017-04-25 (Actual); Status verified 2017-04

CONDITIONS: Stress Disorders, Post-traumatic; Substance Use Disorders
Keywords: peer support; web-based treatment; veterans; PTSD; Substance Use Disorders
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Substance-Related Disorders

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Peer-Supported Web CBT (Experimental): Semi-structured brief sessions conducted weekly for the 12 weeks of study treatment by a certified peer support specialist. Sessions focus on helping participants use the skills they are learning in the Web CBT treatment in their daily lives. Web CBT consists of 24 brief (i.e., 20-minute) modules. Participants will be asked to complete two modules per week. Module topics include The Connection Between PTSD and Substance Use, Motivational Enhancement, Relaxation, Identifying, Evaluating and Challenging Automatic Thoughts, Functional Analyses of Substance Use, Substance Use Refusal Skills, Communication, Anger Management, Pain Management, and Insomnia.
  Interventions: Behavioral: Peer-Supported Web CBT
- Self-Managed Web CBT (Experimental): Self-managed Web CBT consists of 24 brief (i.e., 20-minute) modules. Participants will be asked to complete two modules per week. Module topics include The Connection Between PTSD and Substance Use, Motivational Enhancement, Relaxation, Identifying, Evaluating and Challenging Automatic Thoughts, Functional Analyses of Substance Use, Substance Use Refusal Skills, Communication, Anger Management, Pain Management, and Insomnia.
  Interventions: Behavioral: Self-Managed Web CBT

INTERVENTIONS:
Behavioral: Peer-Supported Web CBT
  Arms: Peer-Supported Web CBT
Behavioral: Self-Managed Web CBT
  Arms: Self-Managed Web CBT

SUMMARY:
Veterans who served in Iraq and Afghanistan have high rates of co-morbid PTSD symptoms and hazardous substance use (HSU). Evidence-based treatments for these problems are available in VA specialty clinics, but multiple barriers lead to low utilization of these treatments. Novel treatment approaches are needed. Previous research supports that 1) primary care-mental health integration (PC-MHI) services are associated with increased treatment engagement, 2) technology-based interventions are well accepted by Veterans and are more effective when delivered with professional support, and 3) Veteran peer services are associated with improved treatment engagement, patient motivation, and overall functioning. This study will add a Peer-Support component to an existing Web-based Cognitive Behavioral Treatment (CBT) for PTSD and HSU called Moving Forward. Preliminary data analyses from our NIAAA-funded trial indicate that participants who used Moving Forward more had larger reductions in PTSD symptoms. Qualitative feedback supports that Veterans want interpersonal interactions while receiving treatment and need help engaging in the treatment more fully. Therefore, this pilot study will investigate if adding peer support to Moving Forward improves patients outcomes. A randomized controlled trial (N=30) comparing Moving Forward to Peer-Supported Moving Forward will be conducted. The peer support component will consist of semi-structured brief sessions conducted weekly for the 12 weeks of study treatment by a VA-certified peer support specialist. Peers will receive study-specific training and weekly supervision from clinicians that are part of the study staff. Primary outcomes will include process outcomes (treatment engagement, patient satisfaction) and clinical outcomes (PTSD symptoms, alcohol and substance use, quality of life).

DETAILED DESCRIPTION:
Veterans who served in Iraq and Afghanistan have high rates of co-morbid PTSD symptoms and hazardous substance use (HSU). Evidence-based treatments for these problems are available in VA specialty clinics, but multiple barriers lead to low utilization of these treatments. Novel treatment approaches are needed. Previous research supports that 1) primary care-mental health integration (PC-MHI) services are associated with increased treatment engagement, 2) technology-based interventions are well accepted by Veterans and are more effective when delivered with professional support, and 3) Veteran peer services are associated with improved treatment engagement, patient motivation, and overall functioning. This study will add a Peer-Support component to an existing Web-based Cognitive Behavioral Treatment (CBT) for PTSD and HSU called Moving Forward. Preliminary data analyses from our NIAAA-funded trial indicate that participants who used Moving Forward more had larger reductions in PTSD symptoms. Qualitative feedback supports that Veterans want interpersonal interactions while receiving treatment and need help engaging in the treatment more fully. Therefore, this pilot study will investigate if adding peer support to Moving Forward improves patients outcomes. A randomized controlled trial (N=30) comparing Moving Forward to Peer-Supported Moving Forward will be conducted. The peer support component will consist of semi-structured brief sessions conducted weekly for the 12 weeks of study treatment by a VA-certified peer support specialist. Peers will receive study-specific training and weekly supervision from clinicians that are part of the study staff. Primary outcomes will include process outcomes (treatment engagement, patient satisfaction) and clinical outcomes (PTSD symptoms, alcohol and substance use, quality of life).

ELIGIBILITY:
Inclusion Criteria:

1. At least 18 years of age,
2. An OEF or OIF or OND veteran (verified via CPRS),
3. Hazardous or harmful substance use as measured by one of the following: a) AUDIT score of >=7 (for women) or >= 8 (for men), b) DAST score of >=2, c) Have exited a controlled environment (e.g., detoxification unit, hospital, or correctional facility) within 30 days of screening AND within 30 days prior to entering the controlled environment report heavy drinking (>3 drinks for women or > 4 drinks for men on 1 or more days) or use of any illegal drugs or misuse of prescription drugs (use in excess of the directions or any non-medical use), 4) Determined to have diagnostic-level PTSD (1 A symptom, 1 B symptom, 3 C symptoms AND 2 D symptoms) or subthreshold PTSD (1 A symptom, 1 B symptom, 3 C symptoms OR 2 D symptoms) on the Clinician Administered PTSD Scale (CAPS),

5) Currently receiving primary medical care at the Syracuse VA Medical Center (verified via CPRS)

Exclusion Criteria:

1. Plans to move out of the area within the next three months,
2. Enrolled in psychotherapy in the last two months focused on substance use or PTSD,
3. Have incurred a change in dose or type of a psychiatric medication that treats PTSD or substance use in the last two months,
4. Inability to understand or provide informed consent,
5. Inability to use English to participate in the consent process, the computerized intervention, or the assessments,
6. In need of alcohol detoxification as determined by a score of > 15 on the Clinical Institute Withdrawal Assessment for Alcohol (CIWA-Ar),
7. Current plan or intent to harm self,
8. Medical chart diagnosis of a current psychotic disorder, including schizophrenia or bi-polar disorder,
9. Cognitive impairment specified by a medical chart diagnosis. Diagnoses include dementia and moderate to severe traumatic brain injury (TBI). Patients with mild TBI were not excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2015-11 (Actual); Primary Completion 2017-04 (Actual); Study Completion 2017-04 (Actual)

PRIMARY OUTCOMES:
PTSD Severity | 12 weeks
  The PTSD Checklist-Specific measures PTSD severity with 17 items rated on a 1-5 scale. Higher numbers indicate greater symptom severity.
Percentage of binge drinking days | 12 weeks
  The Timeline Follow-back measures will record daily alcohol consumption.

CONTACTS AND LOCATIONS:
Overall Officials: Kyle Possemato, Ph.D., Principal Investigator — Syracuse Veterans Affairs Medical Center
Locations (1):
- Syracuse Veterans Affairs Medical Center, Syracuse, New York, United States